CLINICAL TRIAL: NCT03536286
Title: Evaluation to Assess the Asili Intervention in South Kivu, Democratic Republic of Congo
Brief Title: Asili Evaluation in the Democratic Republic of Congo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Refugee Committee (Unknown)
Responsible Party: Principal Investigator, Yvonne (Bonnie) A Maldonado, Chief, Division of Pediatric Infectious Diseases, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 35216
Record Dates: First submitted 2018-04-23; First posted 2018-05-24 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Diarrhea; Cough; Fever; Malnutrition, Child
MeSH Terms: conditions — Diarrhea; Cough; Fever; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: As part of the encouragement intervention, participants (households) will be randomly assigned to the "opportunity" or encouragement arm, where they will be incentivized to participate in the Asili intervention, but are allowed to choose whether or not they actually participate.
  Families will be randomly sampled based on location, and a team of 2 local community champions/data collectors (hired from within the community) will visit each of the encouragement arm homes, supervised by a community outreach liaison. Control households will not receive an individualized home visit.
  Due to numerous factors, including political instability and program implementation delays, our local research team was unable to deploy encouragement as planned.

ARMS (4):
- Encouragement Zone 3 (Experimental): Encouragement households will be randomly sampled based on location, and a team of 2 local community champions/data collectors (hired from within the community) will visit each of the encouragement arm homes. Community champions will be responsible for visiting each home, going door-to-door and speaking with each family individually in order to avoid contamination/cross-over with control households.
  The Asili intervention involves membership into a program; households have the option to opt in or out at any time, without consequence to themselves or the study. The intervention itself involves access to clean water and health clinics. No drugs or medication are administered to individuals through this intervention.
  Interventions: Behavioral: Encouragement
- Control Zone 3 (No Intervention): Control households will still have equal access to the Asili intervention and can gain membership into a program at any time. Regardless of membership status, households have the option to opt in or out at any time, without consequence to themselves or the study. The intervention itself involves access to clean water and health clinics. No drugs or medication are administered to individuals through this intervention.
- Encouragement Zone 4 (Experimental): Encouragement households will be randomly sampled based on location, and a team of 2 local community champions/data collectors (hired from within the community) will visit each of the encouragement arm homes. Community champions will be responsible for visiting each home, going door-to-door and speaking with each family individually in order to avoid contamination/cross-over with control households.
  The Asili intervention involves membership into a program; households have the option to opt in or out at any time, without consequence to themselves or the study. The intervention itself involves access to clean water and health clinics. No drugs or medication are administered to individuals through this intervention.
  Interventions: Behavioral: Encouragement
- Control Zone 4 (No Intervention): Control households will still have equal access to the Asili intervention and can gain membership into a program at any time. Regardless of membership status, households have the option to opt in or out at any time, without consequence to themselves or the study. The intervention itself involves access to clean water and health clinics. No drugs or medication are administered to individuals through this intervention.

INTERVENTIONS:
Behavioral: Encouragement — Households will be visited and encouraged to enroll in Asili
  Arms: Encouragement Zone 3; Encouragement Zone 4

SUMMARY:
The South Kivu province of DRC has experience continuous armed conflict over the last several decades; as a result, livelihoods and health metrics are uniformly poor. Thus, the objective of this study is to determine if an integrated set of social enterprises can improve child health while offering viable and scalable new business opportunities for the community. Specific research questions include the impact of the individual enterprises on (1) child health, (2) access to clean water, and (3) economic opportunities in the region.

DETAILED DESCRIPTION:
The South Kivu province of DRC has experience continuous armed conflict over the last several decades; as a result, livelihoods and health metrics are uniformly poor. Thus, the objective of this study is to determine if an integrated set of social enterprises can improve child health while offering viable and scalable new business opportunities for the community.

Asili ("foundation" in Swahili) is an innovative initiative that aims to implement a suite of social enterprises to provide basic services and employment opportunities in South Kivu, DRC. Asili was co-created by the American Refugee Committee (ARC), an independent non-profit, and IDEO.org using a methodology known as human-centered design (HCD); based on the process, a model of multiple businesses to meet multiple needs was developed, linked under the Asili membership system and coordinated through a centralized database. The Asili model is unique in bringing self-sustaining social enterprises together on a common operational platform to improve both health and economic opportunity in the region. These enterprises are 1) clean water and 2) high quality healthcare clinics.

The team at Stanford University has been recruited as the external evaluator to conduct an impact evaluation of Asili in order to determine whether or not the project goals of reduced child disease as well as increased economic capacity are met. The primary outcome of this impact evaluation study is to determine the effect of the Asili intervention on improving the health of children under five from baseline. Secondary outcomes of this study are to determine the impact of the intervention on enhanced economic activity, food security, and maternal self-esteem and self-efficacy. The investigators hypothesize that under-five children in Asili households will have lower incidence of diarrhea, fever, and cough/short, rapid breathing as well as a higher incidence of vaccination rates.

There is little research on the effects of social enterprise/HCD interventions on health, child health in particular, especially in areas recovering from recent conflict. Therefore, the investigators' aim is to determine if a multi-sectoral approach that can improve livelihoods in DRC can also improve family and child health.

This study will use household surveys at two time points (baseline and endline) to collect information on key indicators from the target populations. For Zones 3 and 4, encouragement design will be used to provide an instrumental variable to analyze the difference in outcomes between the households that enroll in Asili and those that do not. Specific research questions include the impact of the individual enterprises on (1) child health, (2) access to clean water, and (3) economic opportunities in the region.

Encouragement design, a variation on the more commonly known randomized control trial (RCT), is a useful alternative for interventions where it is impractical to require adherence by participants or in situations where offering the intervention to a portion of the population is not possible or ethical. Encouragement involves randomly assigning participants to the "opportunity" or encouragement arm, where efforts are made to motivate participants to take part in an intervention or receive a particular treatment, but are allowed to choose whether or not they actually participate.

Because Asili services will be offered and available to all members of the community and controlling access to services is not possible, encouragement design will be utilized to measure uptake of Asili. Families will be randomly sampled based on location, and a team of 2 local community champions/data collectors (hired from within the community) will visit each of the encouragement arm homes, supervised by a community outreach liaison. Community champions will be responsible for visiting each home, going door-to-door and speaking with each family individually in order to avoid contamination/cross-over with control households.

Champions will spend between 25-45 minutes with members of each household, during which they will explain how Asili works, what the intervention encompasses, and the benefits of joining Asili. The investigators hope to foster a sense of trust in the participants randomized to the encouragement arm by engaging data collectors from the community for these one-on-one exchanges with each household. Control households will also have equal access to Asili services; however, those households will not be visited by community champions individually.

The study populations in the two Zones include families surveyed from the catchment area of the Asili project intervention site in South Kivu. Each of these zones has a population of approximately 10,000 individuals; approximately 850 households were recruited at baseline in each of Zones 3 and 4. Baseline data was completed in Zones 3 and 4 in August 2016 and July 2017, respectively, and follow-up is anticipated in April/May 2018.

ELIGIBILITY:
Inclusion Criteria:

* Living in an Asili catchment area
* Between the age of 18 and 65
* Have at least one child under 5 living at home at baseline
* Able to communicate in the study languages: French, Kiswahili, or Mashi

Exclusion Criteria:

* Suffering from a significant mental deficit, including mental illness, learning difficulties, or substance abuse, which would impair their ability to consent to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9999 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Under-5 child health | up to 15 months
  incidence of diarrhea, fever (as a proxy for malaria), and cough/short, rapid breathing (as a proxy for pneumonia)

SECONDARY OUTCOMES:
Enhanced economic activity | up to 15 months
  Measured through household surveys based on standardized DHS questionnaires; questions include employment and income-generating activities currently undertaken as well as measures of how economic activity within the household has changed after enrolling in Asili
Food security | up to 15 months
  Measured through household surveys based on standardized DHS questionnaires; questions include access to food within the household, number of meals that children have missed, and number of days children have had to go without food.
Vaccination rates | up to 15 months

REFERENCES:
- [Derived] Behl R, Ali S, Altamirano J, Leno A, Maldonado Y, Sarnquist C. Rebuilding child health in South Kivu, Democratic Republic of Congo (DRC): evaluating the Asili social enterprise program. Confl Health. 2022 May 7;16(1):21. doi: 10.1186/s13031-022-00454-0. PMID 35526031